CLINICAL TRIAL: NCT05544981
Title: NITRATE-OCT-CIN Trial: A Randomised, Double-blind, Placebo-controlled Study Investigating the Effects of Dietary Nitrate on Vascular Function, Platelet Reactivity and Restenosis in Stable Angina (Sub-study of the NITRATE-OCT Trial)
Brief Title: NITRATE-OCT-CIN (Sub-Study of NITRATE-OCT)
Acronym: NIT-OCT-CIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17/SC/0020
Record Dates: First submitted 2019-04-09; First posted 2022-09-19 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2022-02

CONDITIONS: Cardiovascular Diseases
Keywords: Stable Angina; Nitrate; Contrast Induced Nephropathy
MeSH Terms: conditions — Cardiovascular Diseases; Angina, Stable

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate-rich beetroot juice (Active Comparator): 70 ml of a beetroot juice concentrate containing ~5 mmol nitrate
  Interventions: Dietary Supplement: Beetroot Juice
- Nitrate-deplete beetroot juice (Placebo Comparator): 70 ml of a beetroot juice concentrate that is nitrate-depleted
  Interventions: Dietary Supplement: Beetroot Juice

INTERVENTIONS:
Dietary Supplement: Beetroot Juice — 70 ml of beetroot juice containing ~5 mmol of inorganic nitrate
  Arms: Nitrate-rich beetroot juice
Dietary Supplement: Beetroot Juice — 70 ml of beetroot juice which is nitrate-depleted
  Arms: Nitrate-deplete beetroot juice

SUMMARY:
The NITRATE-OCT:- Contrast Nephropathy Sub-study is a proof-of concept single center, randomized, clinical trial designed to ascertain whether a dietary NO3- approach might prove useful adjunctive therapy improving renal function and reducing CIN in patients with stable angina undergoing elective angioplasty.

Objectives: To determine whether dietary NO3- ingestion exerts any effect on the glomerular filtration rate (GFR) after the exposure to contrast media.

To determine if dietary NO3- ingestion will decrease the incidence of contrast induced nephropathy.

Setting: The patients will be recruited from an on-going clinical trial NITRATE-OCT. This is a study assessing whether the use of dietary NO3- may reduce the incidence of restenosis following elective angioplasty. This study is recruiting patients with stable angina and single/multiple coronary artery stenosis undergoing elective PCI who are haemodynamically stable (systolic BP>100 mmHg). These patients will be recruited at The Barts Heart Centre at St Bartholomew's Hospital. This is one of the biggest centres in the UK, serving a population of almost two million people from The City of London and The North East up to the M25 and is a 24/7 centre performing approximately 3000 angioplasties a year.

The study will take place in the Clinical Trials Unit, William Harvey Heart Centre.

Target population: A total of 246 patients (male and female, age 18-85) with stable angina as per requirements indicated above. Follow-up will take place in the Clinical Trials Unit, William Harvey Research Institute.

Treatment: Patients will be randomised (using an on line randomisation database) to receive 70 ml of a beetroot juice concentrate containing 4-5 mmol nitrate or nitrate-depleted placebo juice concentrate. This intervention will be taken by the patient daily from one day prior to re-establishment of flow with PCI and stent implantation.

DETAILED DESCRIPTION:
Contrast induced nephropathy (CIN) refers to a form of acute kidney injury (AKI) that occurs after parenteral administration of radio-contrast agent in the absence of other identifiable causes. It is the third most common cause of hospital-acquired renal failure, after decreased renal perfusion and use of nephrotoxic medications. It is generally defined as an increase in serum creatinine concentration of 44 mol/L (0.5 mg/dl) or 25% above baseline within 48 hours after contrast administration. More than 70 years after the first description of a fatal renal function impairment following the use of radiographic contrast media, CIN still represents a major and unmet clinical challenge, as this potential complication is associated with a prolonged hospital stay, a higher hospitalization cost, and a significant increase in morbidity and mortality.

Data suggest that CIN is due to an acute tubular dysfunction, however mechanisms underlying such acute tubular dysfunction in the context of CIN are rather poorly understood. Acute tubular dysfunction seen in settings of CIN is generally less severe and tends to recover more quickly when compared with other forms of acute tubular necrosis. Previous studies have suggested that CIN may be caused by either renal vasoconstriction resulting in medullary hypoxemia or direct cytotoxic injury caused by the contrast agents. Both mechanisms are known to decrease nitric oxide (NO) synthesis and, therefore, may contribute to renal injury. Importantly studies in animal models of contrast induced nephropathy have suggested that decreased levels of NO contributes to this renal injury. Thus the replacement of this 'lost' NO represents an approach that might offer therapeutic benefit.

Patients with chronic renal failure, diabetes mellitus, and heart failure all have a common phenotype of reduced bioavailability of NO, and it is possible that this state accounts for their increased susceptibility to develop contrast media nephrotoxicity. There have been several approaches taken in an attempt to restore NO biovailability in order to prevent development of CIN. N-acetylcysteine has been the most studied, and the most promising compound in this regard. The proposed mechanism of action of N-acetylcysteine is stimulation of NO synthase and increased production of NO. However, in patients with already impaired NO bioavailability due in part to dysfunction of the NO synthase pathways, activation of NO synthase may not generate amounts of sufficient for kidney protection.

A potential solution for elevating endogenous NO levels lies in the chemical reduction of inorganic nitrite (NO2-) to NO. For several decades, NO2- was considered primarily an oxidative product of NO metabolism and possibly a deleterious substance with reputed carcinogenic properties. However, evidence indicates that NO2-, which is abundant in blood and tissues, represents a significant stable intravascular endocrine reservoir and tissue storage form of NO that exerts a number of beneficial effects. Indeed, NO2--derived NO protects against myocardial ischaemia/reperfusion injury in pre-clinical models, protects against experimentally-induced endothelial dysfunction and attenuates platelet reactivity in healthy volunteers and improves endothelial function in hypertensive patients with endothelial dysfunction. In addition, of specific relevance to this project, NO2--derived NO has been shown to be reno-protective in pre-clinical models of renal injury. Since the ingestion of dietary inorganic nitrate (NO3- ) increases endogenous NO levels, the investigators suggest that potential therapeutic benefit could be derived from the use of dietary NO3- in the prevention of CIN.

There is no data assessing the impact of inorganic nitrite/nitrate treatment on CIN in patients undergoing PCI. However, in one small study, post-procedural renal function was compared between 112 patients who received organic nitrates prior to coronary intervention and 87 who did not. Baseline characteristics were similar between the 2 groups. Overall, 43 (21.6%) patients developed CIN post-PCI. Of the patients who received organic nitrates, 15.2% developed renal impairment when compared to 29.9% in those who did not (odds ratio [OR] = 0.42, 95% confidence interval [CI] 0.21-0.84, P = .014). Multivariate logistic regression analysis demonstrated that nitrate use was independently correlated with a reduction in the development of contrast nephropathy (OR = 0.334, 95% CI 0.157-0.709, P = .004). Importantly this study used a single dose of organic nitrate, in part it is likely that this approach was taken due to the major complications with the organic nitrates of the development of tolerance. Indeed, it is this characteristic of these drugs that has profoundly limited their clinical utility. Inorganic dietary nitrate, in contrast, is superior in this respect in that there is no evidence of tolerance with prolonged administration and it possesses a much longer half life (~8 hours) as opposed to minutes with the organic nitrates. The investigators therefore propose to evaluate the effects of dietary NO3- administration on the incidence of CIN in patients undergoing percutaneous coronary intervention.

Specifically with respect to the study of NO2- and CIN; preliminary data from the NITRITE-AMI study performed by the investigators showed that a single bolus of intracoronary NO2- given during primary PCI for ST-elevation MI lead to a significant rise in circulating NO2- levels which lead to a suggestion of reduced CIN. During the first 48 hours after reperfusion, 12.5% of patients in the control group developed CIN, compared to 2.5% patients in the nitrite group (p=0.108). With respect to change in eGFR, from baseline to 48 hours, there was a reduction in eGFR in the placebo group with a trend to an increase in the nitrite group with a significant difference between the change in eGFR over time between the 2 groups (Nitrite group: 5.98 ± 1.99 vs Placebo: -10.15 ±3.69, p=0.002).

Thus, together all of the above issues coupled with preliminary data support the rationale for further exploration of potential approaches based upon elevation of circulating NO2- levels that might reduce the burden of CIN on the NHS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stable angina diagnosed by a cardiologist on optimal medical therapy undergoing angioplasty to treat residual symptoms.
2. Aged 18-85
3. Patients able and willing to give their written informed consent.
4. Patients undergoing successful PCI procedure.

Exclusion Criteria:

1. Unstable ischaemic heart disease, with an episode of chest pain in less than 24 hours.
2. Patients who have had previous coronary artery bypass surgery (CABG), if they are undergoing angioplasty within a non-native vessel.
3. Patients undergoing angioplasty with a bio-absorbable stent.
4. Current diagnosis of or treatment for malignancy, other than non-melanoma skin cancer.
5. Current life-threatening condition other than vascular disease that may prevent a subject completing the study.
6. Use of an investigational device or investigational drug within 30 days or 5 half-lives (whichever is the longer) preceding the first dose of study medication.
7. Patients considered unsuitable to participate by the research team (e.g., due to medical reasons, laboratory abnormalities, or subject's unwillingness to comply with all study related procedures).
8. Severe acute infection, or significant trauma (burns, fractures).
9. Pregnancy. This will be tested by urine HcG measurement
10. History of alcohol or drug abuse within the past 6 months.
11. A history of heart failure NYHA class 3-4 or severe LV dysfunction LVEF<30% regardless of symptom status.
12. Systemic autoimmune disease such as rheumatoid arthritis, connective tissue disease, or other conditions known to be associated with chronic inflammation such as inflammatory bowel disease.
13. Patients who have donated > 500mls blood within 56 days prior to study medication administration.
14. Anaemia with Hb <10g/dl, or any other known blood disorder or significant illness that may affect platelet function, and coagulation.
15. A history of chronic viral hepatitis (including presence of hepatitis B surface antigen or hepatitis C antibody or other chronic hepatic disorder) or HIV.
16. Abnormal liver function due to acute or chronic liver conditions 3 x upper limit of normal at screening.
17. Renal impairment with creatinine clearance (eGFR) of 35ml/min at screening.
18. If patients are on mouthwash, they must be willing to stop using this at least 1 week before the start of the study and throughout the duration that they are involved in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of CIN | 2-3 days post procedure (as Per KDIGO)
  The primary endpoint will be the incidence of CIN (defined as an absolute rise of ≥0.5 mg/dL or a relative increase of ≥25% in serum creatinine over baseline within 48 to 72 h after contrast administration) We will compare the incidence of CIN in patients who received oral nitrate with the of the group that did not receive nitrates.

SECONDARY OUTCOMES:
Change in eGFR from pre to post procedure (within 48hours) | 2 days post procedure
  Difference in real function (eGFR) from baseline to 48hrs
Incidence of Re-hospitalization, haemodialysis and mortality | 6 weeks after contrast admistration
  Adverse events
Plasma levels of NGAL, cystatin-C and measured at 24-72 hours post contrast administration. | 2-3 days post procedure
  Renal biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Jones, MBBS, PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- William Harvey Research Institute, Barts and The London School of Medicine, London, United Kingdom

REFERENCES:
- [Background] Rathod KS, Jones DA, Van-Eijl TJ, Tsang H, Warren H, Hamshere SM, Kapil V, Jain AK, Deaner A, Poulter N, Caulfield MJ, Mathur A, Ahluwalia A. Randomised, double-blind, placebo-controlled study investigating the effects of inorganic nitrate on vascular function, platelet reactivity and restenosis in stable angina: protocol of the NITRATE-OCT study. BMJ Open. 2016 Dec 20;6(12):e012728. doi: 10.1136/bmjopen-2016-012728. PMID 27998900
- [Background] Tripatara P, Patel NS, Webb A, Rathod K, Lecomte FM, Mazzon E, Cuzzocrea S, Yaqoob MM, Ahluwalia A, Thiemermann C. Nitrite-derived nitric oxide protects the rat kidney against ischemia/reperfusion injury in vivo: role for xanthine oxidoreductase. J Am Soc Nephrol. 2007 Feb;18(2):570-80. doi: 10.1681/ASN.2006050450. Epub 2007 Jan 3. PMID 17202421